CLINICAL TRIAL: NCT06940115
Title: Clinical and Radiographical Assessment of Patients With Sub-condylar Fracture Using CAD/CAM Polyetheretherketone (PEEK) Trapezoidal Plates Versus CAD/CAM Titanium Trapezoidal Plates: Randomized Controlled Clinical Study
Brief Title: Clinical and Radiographical Assessment of Patients With Sub-condylar Fracture Using Polyetheretherketone (PEEK) Trapezoidal Plates Versus Titanium Trapezoidal Plates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Yousef Badrasawi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PEEK plate in condyle fracture
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Condylar Neck Fractures; Polyetheretherketone; Mandible Fracture
Keywords: PEEK PLATES; TRAPEZOIDAL PLATES; CAD/CAM
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): CAD/CAM titanium trapezoidal plates
  Interventions: Other: titanium trapezoidal plates
- comparator group (Experimental): CAD/CAM polyetheretherketone (PEEK) trapezoidal plates
  Interventions: Other: PEEK trapezoidal plates

INTERVENTIONS:
Other: titanium trapezoidal plates — ORIF subcondylar fracture using trapezoidal titanium plates
  Arms: control group
Other: PEEK trapezoidal plates — ORIF subcondylar fracture using trapezoidal PEEK plates
  Arms: comparator group

SUMMARY:
Some of titanium's drawbacks that is commonly used in maxillofacial surgery included scatter artefacts on regular imaging, implant exposure and inflammation, high thermal conductivity, and high elastic modulus. Very few clinical studies have been published on using a PEEK plate in the mandibular fractures and to the best of the author's knowledge, this is the first study that will be done comparing trapezoidal condylar 3D printed PEEK plates and titanium trapezoidal condylar plate in subcondylar fractures in terms of clinical and radiographical outcomes.

DETAILED DESCRIPTION:
Mandibular subcondylar fractures are common injuries that require treatment to restore function and aesthetic. Titanium plates have long been the gold standard for fixation in these fractures due to their strength, durability, and ability to provide rigid stabilization. However, they are associated with limitations such as a higher elastic modulus than bone, imaging artifacts (e.g., CT or MRI interference), and hardware-related complications. These drawbacks have prompted interest in alternative materials like polyetheretherketone (PEEK).

PEEK is a novel biomaterial with promising properties, including biocompatibility, a modulus of elasticity closer to bone, and reduced imaging artifacts. These characteristics suggest it may mitigate some of the challenges associated with titanium plates. The improved elasticity of PEEK could reduce stress shielding and enhance functional recovery, while its imaging compatibility could simplify postoperative assessments.

Researchers have shown significant interest in the application of PEEK composites in trauma plating systems, total replacement implants, and tissue scaffolds, highlighting its potential as a versatile biomaterial. Despite these advantages, evidence specifically evaluating PEEK trapezoidal plates for subcondylar fractures remains scarce, there are a no clinical studies directly comparing the outcomes of PEEK and titanium trapezoidal plates in terms of clinical outcomes. Conducting a study to evaluate these two materials would provide valuable evidence to guide material selection in mandibular subcondylar fracture management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, irrespective of gender
* Recent mandibular subcondylar fractures indicated for open reduction and internal fixation

Exclusion Criteria:

* Medically compromised patients contradicting operation (ASA III, IV & V).
* Patients receiving radiotherapy or chemotherapy.
* Infection at the fracture line.
* Pathological fractures and old fractures
* comminuted fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum mouth opening | outcome will be measured postoperatively in 4 different time points. 1st time point is at 1 week after surgery. 2nd time is point at 1 month after surgery. 3rd time point is at 3 months after surgery. 4th time point is at 6 months after surgery
  Maximum mouth opening is the distance between the incisal edges of the upper and lower central incisors at the midline when the mouth is opened as wide as possible without pain. It will be measured in millimeters (mm) using a caliper